CLINICAL TRIAL: NCT00728988
Title: A Prospective Randomized, Open-Label, Parallel-Group Comparative Study: Atorvastatin Pre-Treatment Versus Usual Care In Asian Patients With Acute Coronary Syndromes Undergoing Early Percutaneous Coronary Intervention
Brief Title: Atorvastatin Pre-Treatment Study In Asian Patients With Acute Coronary Syndrome
Acronym: ALPACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A2581161
Record Dates: First submitted 2008-07-31; First posted 2008-08-06 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Asia Lipitor Pre-treatment in Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin Group (Experimental)
  Interventions: Drug: Atorvastatin
- Usual Care Group (Other)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 80mg 12 hours pre-Percutaneous Coronary Intervention (PCI), 40mg 2 hours pre-PCI and 40mg daily after PCI for 30 days.
  Arms: Atorvastatin Group
Drug: Atorvastatin — 40mg daily after PCI for 30 days.
  Arms: Usual Care Group

SUMMARY:
This present study is specifically designed to examine the efficacy and safety of a high pre-treatment dose of atorvastatin in Asian patients with NSTE-ACS in China and the Republic of Korea, by using a treatment paradigm similar to that employed in the ARMYDA-ACS study.

ELIGIBILITY:
Inclusion Criteria:

* Non-ST elevated ACS; LDL-C > 80 mg/dl

Exclusion Criteria:

* ST elevated acute myocardial infarction; previously or currently treated with atorvastatin or other statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- China (7):
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Changsha, Hunan
  - Pfizer Investigational Site, Shenyang, Liaoning
  - Pfizer Investigational Site, Qingdao, Shandong
  - Pfizer Investigational Site, Hangzhou, Zhejiang
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai
- South Korea (10):
  - Pfizer Investigational Site, Seongnam-si, Gyeonggi-do, Korea
  - Pfizer Investigational Site, Busan
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Daejeon
  - Pfizer Investigational Site, Gangneung-si, Gangwon-do
  - Pfizer Investigational Site, Gwangju
  - Pfizer Investigational Site, Jinju-si, Gyeongsangnam-do
  - Pfizer Investigational Site, Koyang-shi
  - Pfizer Investigational Site, Seoul
  - Pfizer Investigational Site, Ulsan

REFERENCES:
- [Derived] Jang Y, Zhu J, Ge J, Kim YJ, Ji C, Lam W. Preloading with atorvastatin before percutaneous coronary intervention in statin-naive Asian patients with non-ST elevation acute coronary syndromes: A randomized study. J Cardiol. 2014 May;63(5):335-43. doi: 10.1016/j.jjcc.2013.09.012. Epub 2013 Nov 9. PMID 24216317
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581161&StudyName=Atorvastatin%20Pre-Treatment%20Study%20In%20Asian%20Patients%20With%20Acute%20Coronary%20Syndrome

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin: Atorvastatin 80 mg 12 hours pre- percutaneous coronary intervention (PCI) and 40 mg 2 hours PCI, and usual care.
- Usual Care: Aspirin 200-300 mg pre-PCI and 100-200 mg daily thereafter; clopidogrel 300 mg loading dose at least 3 hours pre-PCI and 75 mg thereafter; subcutaneous heparin: enoxaparin 1 mg/kg every 12 hours pre-PCI or dalteparin 120 IU/kg every 12 hours pre-PCI; and atorvastatin 40 mg daily after PCI for 30 days.
Period: Overall Study
Arm/Group | Atorvastatin | Usual Care
Started | 247 | 252
Treated | 245 | 250
Full Analysis Set | 163 | 172
Completed | 154 | 164
Not Completed | 93 | 88
Not completed — Not Treated | 2 | 2
Not completed — Death | 1 | 1
Not completed — Adverse Event | 3 | 2
Not completed — Other | 85 | 77
Not completed — Withdrawal by Subject | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Usual Care | Total
Number analyzed (Participants) | 247 | 252 | 499
Age, Customized [Number; unit: participants]
  18 to 44 years | 23 | 9 | 32
  45 to 64 years | 134 | 156 | 290
  >= 65 years | 90 | 87 | 177
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 77 | 158
  Male | 166 | 175 | 341

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Major Adverse Cardiac Events (MACE) (Incidence of MACE) at 30 Days Post-percutaneous Coronary Intervention (PCI)
Description: Percentage calculated as: (number of participants who experienced MACE [death, myocardial infarction, target vessel revascularization] within 30 days post-PCI) divided by (number of participants who experienced PCI) * 100. Major Adverse Cardiac Events (MACE) that occurred after 33 days post PCI were excluded.
Time Frame: 30 days post PCI
Population: Full Analysis Set (FAS): all participants who received at least one dose of study medication and received percutaneous coronary intervention (PCI). Last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin | Usual Care
Number analyzed (Participants) | 163 | 172
percentage of participants
  Total MACE | 14.7 | 15.7
  Death | 0.6 | 0.6
  Myocardial Infarction | 14.1 | 15.1
  Target Vessel Revascularization | 0.0 | 0.0
Statistical Analysis 1: Comparison: Atorvastatin vs Usual Care; Total MACE: treatment difference. Null hypothesis = no difference between the incidence rates in the two groups. A 5% two-sided continuity adjusted Chi-square test was applied; Test type: Superiority or Other; p = 0.9237, Chi-squared, Corrected; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-7.3 to 9.3] — 95% confidence interval for the true difference in the incidence of MACE between the two treatment groups. Difference of incidence = usual care minus atorvastatin
Statistical Analysis 2: Comparison: Atorvastatin vs Usual Care; Death: treatment difference. Null hypothesis = no difference between the incidence rates in two groups. Fisher's exact test was applied because the expected frequency of events was less than 5; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-10.7 to 10.7] — Confidence limits were calculated by the exact unconditional inference. Difference of incidence = usual care minus atorvastatin
Statistical Analysis 3: Comparison: Atorvastatin vs Usual Care; Myocardial Infarction: treatment difference. Null hypothesis = no difference between the incidence rates in the two groups. A 5% two-sided continuity adjusted Chi-square test was applied; Test type: Superiority or Other; p = 0.9158, Chi-squared, Corrected; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-7.2 to 9.2] — Difference of incidence = usual care minus atorvastatin
Statistical Analysis 4: Comparison: Atorvastatin vs Usual Care; Unadjusted odds ratio and 95% confidence interval calculated by including treatment group as the only covariate in the logistic regression model. Reference group = usual care; Test type: Superiority or Other; p = 0.80, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.5104 to 1.6846]
Statistical Analysis 5: Comparison: Atorvastatin vs Usual Care; Adjusted odds ratio: model includes treatment group and potential confounding covariates age, gender, country, non-ST elevation myocardial infarction, LVEF <=40, and use of beta-blockers, ACE-inhibitors, angiotension receptor blockers, calcium channel antagonists, and diuretics. Reference group = usual care; Test type: Superiority or Other; p = 0.90, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.4887 to 1.8836]
Statistical Analysis 6: Comparison: Atorvastatin vs Usual Care; MACE-free survival up to Day 30. A censoring variable with a value of 1 denoted that the subject had the event and 0 indicated that the subject was censored. A log-rank test was applied to investigate any differences on the survival distribution function between two treatment groups; Test type: Superiority or Other; p = 0.8494, Log Rank; Survival analysis: Kaplan-Meier log rank test

2. Secondary Outcome: Percentage of Participants With Major Adverse Cardiac Events (MACE) (Incidence of MACE) at 8 Hours Post-PCI
Description: Percentage calculated as: (number of participants who experienced MACE within 8 hours post-PCI) divided by (number of participants who experienced PCI) * 100.
Time Frame: 8 hours post PCI
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin | Usual Care
Number analyzed (Participants) | 163 | 172
percentage of participants | 6.7 | 6.4
Statistical Analysis 1: Comparison: Atorvastatin vs Usual Care; Treatment difference (%). Null hypothesis = no difference between the incidence rates in the two groups. A 5% two-sided continuity adjusted Chi-square test was applied; Test type: Superiority or Other; p = 1.0000, Chi-squared, Corrected; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-5.6 to 6.3] — Difference of incidence = atorvastatin minus usual care

3. Secondary Outcome: Percentage of Participants With Major Adverse Cardiac Events (MACE) (Incidence of MACE) at 24 Hours Post-PCI
Description: Percentage calculated as: (number of participants who experienced MACE within 24 hours post PCI) divided by (number of participants who experienced PCI) * 100.
Time Frame: 24 hours post PCI
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin | Usual Care
Number analyzed (Participants) | 163 | 172
percentage of participants | 13.5 | 15.1
Statistical Analysis 1: Comparison: Atorvastatin vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7896, Chi-squared, Corrected; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-9.7 to 6.5] — Difference of incidence = atorvastatin minus usual care

4. Secondary Outcome: Percentage of Participants With Elevated Creatine Kinase-MB (CK-MB)
Description: CK-MB above the upper limit of normal range from baseline (biomarker of myocardial injury); normal range: 0-5.0 nanograms per milliliter (ng/mL).
Time Frame: 8 hours, 24 hours and 30 days post PCI
Population: FAS. N = number of participants with baseline and at least one post-baseline response.
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin | Usual Care
Number analyzed (Participants) | 160 | 169
percentage of participants
  8 Hours Post-PCI | 11.3 | 13.6
  24 Hours Post-PCI | 15.6 | 18.9
  30 Days Post-PCI | 1.3 | 0.0
Statistical Analysis 1: Comparison: Atorvastatin vs Usual Care; 8 hours post-PCI: difference (%) in proportions. Null hypothesis = no difference in proportions of the two groups. A 5% two-sided continuity adjusted Chi-square test was applied; Test type: Superiority or Other; p = 0.631, Chi-squared, Corrected; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-10.1 to 5.4]
Statistical Analysis 2: Comparison: Atorvastatin vs Usual Care; 24 hours post-PCI: difference (%) in proportions. Null hypothesis = no difference in proportions of the two groups. A 5% two-sided continuity adjusted Chi-square test was applied; Test type: Superiority or Other; p = 0.518, Chi-squared, Corrected; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-12.1 to 5.5]
Statistical Analysis 3: Comparison: Atorvastatin vs Usual Care; 30 days post-PCI: difference (%) in proportions. Null hypothesis = no difference in proportions of the two groups. Fisher's exact test was applied because the expected frequency of biomarker elevation was less than 5; Test type: Superiority or Other; p = 0.236, Fisher Exact; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-9.6 to 12.0]

5. Secondary Outcome: Percentage of Participants With Elevated Troponin I
Description: Troponin I above the upper limit of normal range from baseline (biomarker of myocardial injury): normal range: 0-0.5 nanograms per milliliter (ng/mL).
Time Frame: 8 hours, 24 hours and 30 days post PCI
Population: FAS. N = number of participants with baseline and at least one post-baseline response.
Measure: Number; unit: percentage of participants
Groups:
- Atorvastatin: Atorvastatin 80 mg 12 hours pre-PCI and 40 mg 2 hours pre-percutaneous coronary intervention (PCI), and usual care.
Arm/Group | Atorvastatin | Usual Care
Number analyzed (Participants) | 161 | 169
percentage of participants
  8 hours post-PCI | 40.4 | 35.5
  24 hours post-PCI | 49.7 | 44.4
  30 days post-PCI | 1.9 | 1.8
Statistical Analysis 1: Comparison: Atorvastatin vs Usual Care; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.425, Chi-squared, Corrected; Mean Difference (Final Values) = 4.9, 95% CI 2-sided [-6.2 to 15.9]
Statistical Analysis 2: Comparison: Atorvastatin vs Usual Care; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.392, Chi-squared, Corrected; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [-6.1 to 16.7]
Statistical Analysis 3: Comparison: Atorvastatin vs Usual Care; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 1.000, Fisher Exact; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-10.7 to 10.9]

6. Secondary Outcome: Percentage of Participants With Elevated Myoglobin
Description: Myoglobin above the upper limit of normal from baseline (biomarker of myocardial injury): normal range: 0-109 nanograms per milliliter (ng/mL).
Time Frame: 8 hours, 24 hours and 30 days post PCI
Population: FAS. N = number of participants with baseline and at least one post-baseline response.
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin | Usual Care
Number analyzed (Participants) | 159 | 166
percentage of participants
  8 hours post-PCI | 8.2 | 10.8
  24 hours post-PCI | 3.1 | 4.2
  30 days post-PCI | 1.3 | 0.6
Statistical Analysis 1: Comparison: Atorvastatin vs Usual Care; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.529, Chi-squared, Corrected; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-9.6 to 4.3]
Statistical Analysis 2: Comparison: Atorvastatin vs Usual Care; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.827, Chi-squared, Corrected; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-5.8 to 3.6]
Statistical Analysis 3: Comparison: Atorvastatin vs Usual Care; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.616, Fisher Exact; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-10.3 to 11.5]

7. Secondary Outcome: Percent Change From Baseline in C-Reactive Protein (CRP)
Description: C-reactive protein percent change from baseline = (post baseline value minus baseline value) divided by baseline value*100. Includes all CRP samples tested for the study, including samples unaffected and those samples affected by defective high-sensitivity (hs) CRP reagents.
Time Frame: Baseline, 8 hours, 24 hours and 30 days
Population: FAS. N = number of subjects with non-missing values at baseline.
Measure: Least Squares Mean (Standard Error); unit: percent change in CRP
Arm/Group | Atorvastatin | Usual Care
Number analyzed (Participants) | 161 | 169
percent change in CRP
  8 hours post-PCI | 205.25 (67.799) | 234.77 (66.135)
  24 hours post-PCI | 594.07 (110.774) | 543.50 (107.730)
  30 days post-PCI | 9.01 (58.276) | 67.23 (56.562)
Statistical Analysis 1: Comparison: Atorvastatin vs Usual Care; 8 hours post-PCI: difference (% change); Test type: Superiority or Other; p = 0.7554, ANOVA; Mean Difference (Final Values) = -29.53, 95% CI 2-sided [-215.87 to 156.81]
Statistical Analysis 2: Comparison: Atorvastatin vs Usual Care; 24 hours post-PCI: difference (% change); Test type: Superiority or Other; p = 0.7436, ANOVA; Mean Difference (Final Values) = 50.58, 95% CI 2-sided [-253.42 to 354.58]
Statistical Analysis 3: Comparison: Atorvastatin vs Usual Care; 30 days post-PCI: difference (% change); Test type: Superiority or Other; p = 0.4741, ANOVA; Mean Difference (Final Values) = -58.22, 95% CI 2-sided [-218.12 to 101.68]

ADVERSE EVENTS:
Description: Safety analysis set: all randomized subjects with at least 1 dose of treatment. An adverse event (AE) term may be reported as both a serious and a non-serious AE, but are distinct events. AE may = serious for 1 subject and non-serious for another subject, or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Atorvastatin | Usual Care
Serious Adverse Events (participants affected / at risk) | 16/245 | 16/250
Other Adverse Events (participants affected / at risk) | 65/245 | 45/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=245) | Usual Care (N=250)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 4
Palpitations (Cardiac disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 4 | 7
Alanine aminotransferase increased (Investigations) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=245) | Usual Care (N=250)
Myocardial infarction (Cardiac disorders) | 15 | 12
Chest pain (General disorders) | 13 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 7
Headache (Nervous system disorders) | 29 | 18

LIMITATIONS AND CAVEATS:
Defective high-sensitivity C reactive protein reagents showed instability and 20% average positive bias in results, affecting only change from baseline in CRP. Analyses were performed on all samples; results include affected and unaffected samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.